CLINICAL TRIAL: NCT02493881
Title: Descriptive in Vivo Study of Evaluating the Motor Function of Recurrent Laryngeal Nerve's Extralaryngeal Branching Electromyographically.
Brief Title: Recurrent Laryngeal Nerve's Motor Function: Sometimes Motor Fibers May Also Be Located in The Posterior Branch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Uludag, Associated Professor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SEEAH01
Record Dates: First submitted 2015-06-26; First posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Recurrent Laryngeal Nerve Injuries
Keywords: Motor function of the extralaryngeal branches; intraoperative neuromonitoring; recurrent laryngeal nerve
MeSH Terms: conditions — Recurrent Laryngeal Nerve Injuries | interventions — Intraoperative Neurophysiological Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): The RLNs having motor function on the anterior branch assessed by intraoperative neuromonitoring.
  Interventions: Device: intraoperative neuromonitoring
- Group 2 (Active Comparator): RLNs having motor function on anterior and posterior branch assessed by intraoperative neuromonitoring.
  Interventions: Device: intraoperative neuromonitoring

INTERVENTIONS:
Device: intraoperative neuromonitoring — NIM-Response 3.0 Intraoperative Neuromonitoring System (Medtronic Xomed, Jacksonville, FL, USA) was used to record the EMG amplitude signal for the anterior and/or posterior branches of recurrent laryngeal nerves (RLNs).

SUMMARY:
The investigators hypothesized that, sometimes the posterior branch of the recurrent laryngeal nerve may also have motor function. The investigators aimed to evaluate motor function of the branches in the branching recurrent laryngeal nerves in this study.

DETAILED DESCRIPTION:
This study group consisted of consecutive patients, undergoing thyroid and parathyroid surgery with IONM. Both anterior and posterior branches of the recurrent laryngeal nerves were assessed separately by both electromyography endotracheal tube for adduction and finger palpation for detection of laryngeal twitch due to posterior cricoarytenoid abduction. The recurrent laryngeal nerves having motor function only in the anterior branches were defined as group 1, whereas the nerves having motor function both in the anterior and posterior branches were as group 2.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent parathyroid/thyroid surgery with intraoperative neuromonitoring ,
2. Patients who had normal vocal cord functions preoperatively. -

Exclusion Criteria:

1. Preoperative recurrent laryngeal nerve palsy,
2. Intentional nerve transection because of cancer invasion,
3. Assessment failure of recurrent laryngeal nerve function due to the deficiency of the intraoperative neuromonitoring equipment,.
4. Parathyroidectomy operations that recurrent laryngeal nerves were not fully dissected.

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The evoked EMG potentials of the branches of the recurrent laryngeal nerves as microvolt, by intraoperative neuromonitoring. | intraoperative
  The nerves , due to having motor functions whether on their anterior or posterior branches, were divided into two groups. The amplitudes of the anterior and posterior branches within the group 2 were compared.

SECONDARY OUTCOMES:
The diameters of the branches of the recurrent laryngeal nerves. | intraoperative
  The branch diameters of the recurrent laryngeal nerves were compared between the two groups.
The branching distances of the recurrent laryngeal nerves. | intraoperative
  The branching distances of the recurrent laryngeal nerves till the entry point into the larynx, were compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Isgor, Prof., Study Director — Bahcesehir University Medical Faculty, Department of General Surgery

REFERENCES:
- [Result] Gurleyik E. Location of motor fibers within branches of the recurrent laryngeal nerve with extralaryngeal terminal bifurcation; Functional identification by intraoperative neuromonitoring. Surgery. 2015 Nov;158(5):1339-44. doi: 10.1016/j.surg.2015.04.019. Epub 2015 Jun 6. PMID 26054316
- [Result] Fontenot TE, Randolph GW, Friedlander PL, Masoodi H, Yola IM, Kandil E. Gender, race, and electrophysiologic characteristics of the branched recurrent laryngeal nerve. Laryngoscope. 2014 Oct;124(10):2433-7. doi: 10.1002/lary.24631. Epub 2014 Mar 25. PMID 24493270
- [Result] Serpell JW, Yeung MJ, Grodski S. The motor fibers of the recurrent laryngeal nerve are located in the anterior extralaryngeal branch. Ann Surg. 2009 Apr;249(4):648-52. doi: 10.1097/SLA.0b013e31819ed9a4. PMID 19300223
- [Result] Chiang FY, Lu IC, Chen HC, Chen HY, Tsai CJ, Hsiao PJ, Lee KW, Wu CW. Anatomical variations of recurrent laryngeal nerve during thyroid surgery: how to identify and handle the variations with intraoperative neuromonitoring. Kaohsiung J Med Sci. 2010 Nov;26(11):575-83. doi: 10.1016/S1607-551X(10)70089-9. PMID 21126710
- [Result] Cernea CR, Hojaij FC, De Carlucci D Jr, Gotoda R, Plopper C, Vanderlei F, Brandao LG. Recurrent laryngeal nerve: a plexus rather than a nerve? Arch Otolaryngol Head Neck Surg. 2009 Nov;135(11):1098-102. doi: 10.1001/archoto.2009.151. PMID 19917921
- [Result] Casella C, Pata G, Nascimbeni R, Mittempergher F, Salerni B. Does extralaryngeal branching have an impact on the rate of postoperative transient or permanent recurrent laryngeal nerve palsy? World J Surg. 2009 Feb;33(2):261-5. doi: 10.1007/s00268-008-9832-1. PMID 19023612
- [Result] Kandil E, Abdel Khalek M, Aslam R, Friedlander P, Bellows CF, Slakey D. Recurrent laryngeal nerve: significance of the anterior extralaryngeal branch. Surgery. 2011 Jun;149(6):820-4. doi: 10.1016/j.surg.2011.02.012. Epub 2011 Apr 17. PMID 21497872
- [Result] Kandil E, Abdelghani S, Friedlander P, Alrasheedi S, Tufano RP, Bellows CF, Slakey D. Motor and sensory branching of the recurrent laryngeal nerve in thyroid surgery. Surgery. 2011 Dec;150(6):1222-7. doi: 10.1016/j.surg.2011.09.002. PMID 22136844